CLINICAL TRIAL: NCT05788237
Title: A Study to Evaluate the Safety, Tolerability, and Immunogenicity of Respiratory Combination Vaccine Candidates in Older Adults
Brief Title: A Study to Examine Respiratory Combination Vaccines Against Respiratory Syncytial Virus (RSV) and Flu in Older Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: C5401001
Record Dates: First submitted 2023-03-03; First posted 2023-03-28 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Flu; Influenza; Vaccine; RNA vaccine; RSV; Respiratory Syncytial Virus; Combination vaccine; Vaccine osmolality
MeSH Terms: conditions — Influenza, Human | interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: Substudy A: Approximately 250 healthy adults ≥60 years of age will be randomized 1:1 to either Group 1: combination (RSVpreF + qIRV) (Visit 1) followed by placebo (Visit 2); or Group 2: sequential administration of qIRV (Visit 1) followed by RSVpreF (Visit 2) administered 1 month apart. Randomization will be stratified by 3 age groups (60-64, 65-79, and ≥80 years) within each study site.
  Substudy B: Approximately 200 healthy adults ≥50 years of age will be randomized 1:1 to either Group 1: combination (RSVpreF + qIRV) 1.0-mL formulation; or Group 2: combination (RSVpreF + qIRV) 0.5 mL formulation. Randomization will be stratified by 6 age/sex groups (female 50-64, female 65-79, and female ≥80 years; male 50-64, male 65-79, and male ≥80 years) within the study site.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Substudy A: This is an observer-blinded study. Participants will be blinded to their assigned study intervention. The study staff receiving, storing, dispensing, preparing, and administering the study interventions will be unblinded. All other study and site personnel, including the investigator and investigator staff, will be blinded to assignment of study intervention.
  With the exception of the staff conducting the immunogenicity assays, the sponsor will be unblinded.
  Substudy B: This is an observer-blinded study. Participants will be blinded to their assigned study intervention. The study staff receiving, storing, dispensing, preparing, and administering the study interventions will be unblinded. All other study and site personnel, including the investigator and investigator staff, will be blinded to assignment of study intervention.
  With the exception of the staff conducting the immunogenicity assays, the sponsor will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- SSA Group 1: Combination (Experimental): Combination (RSVpreF + qIRV) (Visit 1) followed by placebo (Visit 2). RSVpreF and qIRV are administered as concomitantly but as individual injections.
  Interventions: Biological: RSVpreF+qIRV; Drug: Placebo
- SSA Group 2: Sequential (Experimental): Sequential administration of qIRV (Visit 1) followed by RSVpreF (Visit 2)
  Interventions: Biological: qIRV; Biological: RSVpreF
- SSB Group 1: Combination (RSVpreF + qIRV) 1.0-mL formulation (Experimental): RSVpreF lyophilized cake reconstituted with water for injection and mixed with qIRV, yielding an injection volume of 1.0 mL
  Interventions: Biological: RSVpreF + qIRV 1.0 mL formulation
- SSB Group 2: Combination (RSVpreF +qIRV) 0.5-mL formulation (Experimental): RSVpreF lyophilized cake reconstituted with qIRV to yield an injection volume of 0.5 mL
  Interventions: Biological: RSVpreF + qIRV 1.0 mL formulation; Biological: RSVpreF + qIRV 0.5 mL formulation

INTERVENTIONS:
Biological: RSVpreF+qIRV — RSVpreF containing 2 stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B combined with Quadrivalent influenza modRNA vaccine (qIRV) encoding HA of 4 strains as recommended for the influenza season (2 A strains, 2 B strains)
  Arms: SSA Group 1: Combination
Biological: qIRV — Quadrivalent influenza modRNA vaccine (qIRV) encoding HA of 4 strains as recommended for the influenza season (2 A strains, 2 B strains)
  Other Names: PF-07252220
  Arms: SSA Group 2: Sequential
Biological: RSVpreF — RSVpreF containing 2 stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B
  Other Names: PF-06928316
  Arms: SSA Group 2: Sequential
Drug: Placebo — 0.9% saline for injection
  Arms: SSA Group 1: Combination
Biological: RSVpreF + qIRV 1.0 mL formulation — RSVpreF containing 2 Stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B plus qIRV Encoding HA of 4 strains as recommended for the influenza season (2 A strains and 2 B strains) plus sterile water as diluent for injection
  Other Names: PF-07941314
  Arms: SSB Group 1: Combination (RSVpreF + qIRV) 1.0-mL formulation; SSB Group 2: Combination (RSVpreF +qIRV) 0.5-mL formulation
Biological: RSVpreF + qIRV 0.5 mL formulation — RSVpreF containing 2 Stabilized RSV prefusion F antigens, in equal amounts from virus subgroups A and B plus qIRV Encoding HA of 4 strains as recommended for the influenza season (2 A strains and 2 B strains)
  Other Names: PF-07941314
  Arms: SSB Group 2: Combination (RSVpreF +qIRV) 0.5-mL formulation

SUMMARY:
Substudy A: The study aims to learn about the safety and effects of two new vaccines for RSV (RSVpreF) and influenza (modRNA qIRV) when given as a single shot compared to when given separately. RSV and influenza lead to infections, mainly in the fall and winter. These vaccines are being developed to help prevent respiratory syncytial virus (RSV) and influenza (Flu) disease.

This study is seeking participants who:

* are 60 years or older
* are healthy or have well-controlled chronic conditions
* have not had a flu shot in the last 120 days
* and agree to be present for all study visits, procedures, and blood draws.

The participants will be divided into 2 groups. Group 1 will receive RSVpreF plus qIRV combo shot, after which participants will receive the placebo (a shot which has no medicine). Group 2 will receive shots for qIRV first and then RSVpreF 1 month apart.

The investigators will examine the experiences of the participants receiving the study vaccines. This will help the investigators determine if the study vaccines are safe and produce a similar immune response.

Participants will be involved in this study for 2 months. During this time, participants will have 3 visits at the study clinic.

Substudy B will investigate 2 formulations of RSVpreF + qIRV of different volumes and osmolaities (concentrations). These formulations will be examined for safety, tolerability, and immunogenicity, with the goal of selecting a formulation for further study.

This study is seeking participants who:

* are 50 years or older
* are healthy or have well-controlled chronic conditions
* have not had a flu shot in the last 180 days
* and agree to be present for all study visits, procedures, and blood draws.

The participants will be divided into 2 groups. Group 1 will receive RSVpreF plus qIRV in a 1.0-mL formulation while Group 2 will receive RSVpreF plus qIRV in a 0.5-mL formulation.

The investigators will examine the experiences of the participants receiving the study vaccines. This will help the investigators determine if the study vaccines are safe, well tolerated and produce a similar immune response.

Participants will be involved in this study for 1 month. During this time, participants will have 2 visits at the study clinic.

DETAILED DESCRIPTION:
Substudy A: This study is designed to evaluate the safety, tolerability, and immunogenicity of respiratory combination vaccine candidates. This initial study will be conducted as a Phase 1b, parallel-group, randomized, placebo-controlled, observer-blinded substudy of RSVpreF and a nucleoside-modified RNA vaccine (qIRV) against RSV and influenza when administered as a combined vaccine and when administered alone.

Healthy adults ≥60 years of age will be randomized 1:1 to either Group 1: combination (RSVpreF + qIRV) followed by placebo; or Group 2: sequential administration of qIRV followed by RSVpreF administered 1 month apart.

Substudy B will be conducted as a Phase 1b, parallel-group, randomized, observer-blinded substudy of RSVpreF and a nucleoside-modified RNA vaccine (qIRV) against RSV and influenza administered as a combined vaccine in a 1.0-mL formulation and when administered in a 0.5-mL formulation.

Healthy adults ≥50 years of age will be randomized 1:1 to either Group 1: combination (RSVpreF + qIRV) 1.0-mL formulation; or Group 2: combination (RSVpreF + qIRV) 0.5 mL formulation. Approximately 100 participants will be randomized within the 50- through 64-year-old group, and 100 participants ≥65 years of age will be randomized.

ELIGIBILITY:
Substudy A:

Inclusion Criteria:

1. Participants ≥60 years of age at study enrollment.
2. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
4. Capable of giving and having signed the informed consent as described in the protocol, which includes complying with the requirements and restrictions listed in the ICD and in this protocol.
5. Receipt of licensed influenza vaccination for the 2022-2023 northern hemisphere season or 2022 southern hemisphere season >120 days before study intervention administration.

Exclusion Criteria:

1. A confirmed diagnosis of RSV infection or influenza ≤120 days before study intervention administration.
2. History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
3. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate IM injection.
4. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before study intervention administration, or planned receipt throughout the study.
8. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration, or planned receipt throughout the study.
9. Receipt of any licensed RSV vaccine at any time prior to enrollment, or planned receipt throughout the study.
10. Receipt of any licensed influenza vaccine ≤120 days before study enrollment, or planned receipt throughout the study.
11. Participation in other studies involving an investigational RSV or mRNA influenza vaccine at any time prior to enrollment, and thereafter until study completion, regardless of vaccine assignment.
12. Participation in any other interventional studies within 28 days before study enrollment through study completion.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Substudy B

Inclusion Criteria:

1. Participants ≥50 years of age at study enrollment.
2. Participants who are willing and able to comply with all scheduled visits, investigational plan, laboratory tests, lifestyle considerations, and other study procedures.
3. Healthy participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion in the study.
4. Capable of giving and having signed the informed consent as described in the protocol, which includes complying with the requirements and restrictions listed in the ICD and in this protocol.
5. Receipt of licensed influenza vaccination for the 2022-2023 northern hemisphere season or 2022 southern hemisphere season >180 days before study intervention administration.

Exclusion Criteria:

1. A confirmed diagnosis of RSV infection or influenza ≤120 days before study intervention administration.
2. History of severe adverse reaction associated with any vaccine and/or severe allergic reaction (eg, anaphylaxis) to any component of the study intervention(s).
3. Bleeding diathesis or condition associated with prolonged bleeding that would, in the opinion of the investigator, contraindicate IM injection.
4. Serious chronic disorder, including metastatic malignancy, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the participant from participating in the study.
5. Immunocompromised individuals with known or suspected immunodeficiency, as determined by history and/or laboratory/physical examination.
6. Other medical or psychiatric condition including recent (within the past year) or active suicidal ideation/behavior or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
7. Receipt of chronic systemic treatment with known immunosuppressant medications (including cytotoxic agents or systemic corticosteroids), or radiotherapy, within 60 days before study intervention administration, or planned receipt throughout the study.
8. Receipt of blood/plasma products or immunoglobulin, from 60 days before study intervention administration, or planned receipt throughout the study.
9. Receipt of any RSV vaccine at any time prior to enrollment, or planned receipt throughout the study.
10. Receipt of any influenza vaccine ≤180 days before study enrollment, or planned receipt throughout the study.
11. Participation in other studies involving an investigational RSV vaccine or mRNA influenza vaccine at any time prior to enrollment, and thereafter until study completion, regardless of vaccine assignment.
12. Participation in any other interventional studies within 28 days before study enrollment through study completion. Participation in purely observational studies is acceptable.
13. Investigator site staff directly involved in the conduct of the study and their family members, site staff otherwise supervised by the investigator, and sponsor and sponsor delegate employees directly involved in the conduct of the study and their family members.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 508 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Hospital Militar Central Cirujano Mayor Dr. Cosme Argerich, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5401001

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had sub-study A (SSA) and sub-study B (SSB).
Pre-assignment Details: A total of 508 participants (SSA: 273 + SSB: 235) were enrolled in this study, 455 participants (SSA:251 + SSB: 204) were randomized to receive study intervention.
Groups:
- SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo: Participants aged >= 60 years were randomized to receive 1.0 mL combination of RSVpreF and qIRV intramuscularly on Day 1 [Vaccination 1]. After 1 month, placebo (0.9% normal saline for injection) [Vaccination 2] was administered intramuscularly. Participants were followed up to maximum of 35 days after Vaccination 2.
- SSA: Group 2: Sequential Administration qIRV/ RSVpreF: Participants aged >= 60 years were randomized to receive 1.0 mL of qIRV intramuscularly on Day 1 (Vaccination 1). After 1 month, RSVpreF (Vaccination 2) was administered intramuscularly. Participants were followed up to maximum of 35 days after Vaccination 2.
- SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation: Participants aged >=50 years were randomized to receive 1.0 mL of combination of RSVpreF and qIRV intramuscularly on Day 1. Participants were followed up to maximum of 35 days after Vaccination.
- SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation: Participants aged >=50 years were randomized to receive 0.5 mL of combination of RSVpreF and qIRV intramuscularly on Day 1. Participants were followed up to maximum of 35 days after Vaccination.
Period: SSA (Approximately 2 Months)
Arm/Group | SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo | SSA: Group 2: Sequential Administration qIRV/ RSVpreF | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Started | 125 | 126 | 0 (Participants of SSB did not enter SSA. Period only for SSA, hence no participants for SSB.) | 0 (Participants of SSB did not enter SSA. Period only for SSA, hence no participants for SSB.)
Vaccination 1 | 125 ((RSVpreF + qIRV)) | 126 ((qIRV)) | 0 | 0
Vaccination 2 | 121 ((Placebo)) | 116 ((RSVpreF)) | 0 | 0
Completed | 120 | 113 | 0 | 0
Not Completed | 5 | 13 | 0 | 0
Not completed — No longer met eligibility criteria | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 8 | 0 | 0
Not completed — Adverse Event | 1 | 2 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: SSB (Approximately 1 Month)
Arm/Group | SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo | SSA: Group 2: Sequential Administration qIRV/ RSVpreF | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Started | 0 (Participants of SSA did not enter SSB. Period only for SSB, hence no participants for SSA.) | 0 (Participants of SSA did not enter SSB. Period only for SSB, hence no participants for SSA.) | 102 | 102
Vaccination | 0 | 0 | 101 | 102
Completed | 0 | 0 | 101 | 100
Not Completed | 0 | 0 | 1 | 2
Not completed — Not Vaccinated | 0 | 0 | 1 | 0
Not completed — Refused further study procedures | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population was evaluated. SSA= All enrolled participants who received the study intervention either in combination RSVpreF + qIRV, or as placebo, qIRV, or RSVpreF alone. SSB= All enrolled participants who received the study intervention (0.5 mL or 1.0 mL).
Groups:
- Total: Total of all reporting groups
Arm/Group | SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo | SSA: Group 2: Sequential Administration qIRV/ RSVpreF | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation | Total
Number analyzed (Participants) | 125 | 126 | 101 | 102 | 454
Age, Customized [Count of Participants; unit: Participants]
  50-64 years | 22 | 23 | 50 | 52 | 147
  65-79 years | 94 | 93 | 48 | 47 | 282
  >=80 years | 9 | 10 | 3 | 3 | 25
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 73 | 47 | 48 | 230
  Male | 63 | 53 | 54 | 54 | 224
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 125 | 126 | 101 | 101 | 453
  Not Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 125 | 126 | 101 | 102 | 454
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: SSA: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 1
Description: Local reactions included pain, redness and swelling at the injection site, recorded by participants in an electronic diary (e-diary). Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity; severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as mild: 2.5 cm to 5.0 cm; moderate: greater than (>) 5.0 cm to 10.0 cm; severe: > 10 cm.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination 1
Population: SSA: E-diary safety population consisted of all enrolled participants who received the study intervention either in combination RSVpreF + qIRV, or as placebo, qIRV, or RSVpreF alone, and had at least 1 day of e-diary data transferred.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: Group 1: RSVpreF + qIRV: Participants received 1 mL of combination of RSVpreF and qIRV intramuscularly on Day 1 [Vaccination 1].
- SSA: Group 2: qIRV: Participants received 1 mL of qIRV intramuscularly on Day 1 [Vaccination 1].
Arm/Group | SSA: Group 1: RSVpreF + qIRV | SSA: Group 2: qIRV
Number analyzed (Participants) | 125 | 125
Percentage of participants
  Pain at the injection site: Mild | 49.6 [40.5 to 58.7] | 52.0 [42.9 to 61.0]
  Pain at the injection site: Moderate | 20.8 [14.1 to 29.0] | 28.0 [20.3 to 36.7]
  Pain at the injection site: Severe | 0 [0.0 to 2.9] | 2.4 [0.5 to 6.9]
  Redness: Mild | 3.2 [0.9 to 8.0] | 3.2 [0.9 to 8.0]
  Redness: Moderate | 4.0 [1.3 to 9.1] | 4.8 [1.8 to 10.2]
  Redness: Severe | 0 [0.0 to 2.9] | 0.8 [0.0 to 4.4]
  Swelling: Mild | 5.6 [2.3 to 11.2] | 6.4 [2.8 to 12.2]
  Swelling: Moderate | 3.2 [0.9 to 8.0] | 8.0 [3.9 to 14.2]
  Swelling: Severe | 0.8 [0.0 to 4.4] | 2.4 [0.5 to 6.9]

2. Primary Outcome: SSA: Percentage of Participants With Local Reactions Within 7 Days After Vaccination 2
Description: Local reactions included pain, redness and swelling at the injection site, recorded by participants in an e-diary. Pain at injection site was graded as mild: did not interfere with activity; moderate: interfered with activity; severe: prevented daily activity. Redness and swelling were measured and recorded in measuring device units, where 1 measuring device unit=0.5 cm. Redness and swelling were graded as mild: 2.5 cm to 5.0 cm; moderate: > 5.0 cm to 10.0 cm; severe: > 10 cm.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination 2 (1 Month After Vaccination 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: Group 1: Placebo: Participants received placebo intramuscularly on 1 month after Vaccination 1 [Vaccination 2].
- SSA: Group 2: RSVpreF: Participants received 1 mL of RSVpreF intramuscularly on 1 month after Vaccination 1 [Vaccination 2].
Arm/Group | SSA: Group 1: Placebo | SSA: Group 2: RSVpreF
Number analyzed (Participants) | 121 | 115
Percentage of participants
  Pain at the injection site: Mild | 1.7 [0.2 to 5.8] | 7.8 [3.6 to 14.3]
  Pain at the injection site: Moderate | 1.7 [0.2 to 5.8] | 0.9 [0.0 to 4.7]
  Pain at the injection site: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Redness: Mild | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Redness: Moderate | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Redness: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Swelling: Mild | 0.8 [0.0 to 4.5] | 0.9 [0.0 to 4.7]
  Swelling: Moderate | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Swelling: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]

3. Primary Outcome: SSB: Percentage of Participants With Local Reactions Within 7 Days After Vaccination
Description: as for outcome 2
Time Frame: SSB: From Day 1 to Day 7 after Vaccination
Population: SSB: E-diary safety population consisted of all enrolled participants who received the study intervention (0.5 mL or 1.0 mL) and with at least 1 day of e-diary data transferred.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation: Participants aged >=50 years received 1.0 mL of combination of RSVpreF and qIRV intramuscularly on Day 1. Participants were followed up to maximum of 35 days after Vaccination.
- SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation: Participants aged >=50 years received 0.5 mL of combination of RSVpreF and qIRV intramuscularly on Day 1. Participants were followed up to maximum of 35 days after Vaccination.
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 101 | 102
Percentage of participants
  Pain at the injection site: Mild | 42.6 [32.8 to 52.8] | 43.1 [33.4 to 53.3]
  Pain at the injection site: Moderate | 31.7 [22.8 to 41.7] | 32.4 [23.4 to 42.3]
  Pain at the injection site: Severe | 1.0 [0.0 to 5.4] | 2.9 [0.6 to 8.4]
  Redness: Mild | 2.0 [0.2 to 7.0] | 2.0 [0.2 to 6.9]
  Redness: Moderate | 0 [0.0 to 3.6] | 3.9 [1.1 to 9.7]
  Redness: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]
  Swelling: Mild | 4.0 [1.1 to 9.8] | 5.9 [2.2 to 12.4]
  Swelling: Moderate | 5.9 [2.2 to 12.5] | 7.8 [3.4 to 14.9]
  Swelling: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]

4. Primary Outcome: SSA: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, fatigue, headache, vomiting, nausea, diarrhea, chills, new/worsened muscle pain and new/worsened joint pain. These were recorded by participants in an e-diary. Fever defined as oral temperature >=38.0 degrees Celsius (deg C) and categorized as mild: >=38.0 to 38.4 deg C, moderate: >38.4 to 38.9 deg C, severe: >38.9 to 40.0 deg C. Vomiting categorized as mild: 1-2 times in 24 hours (h); moderate: >2 times in 24h; severe: required intravenous (IV) hydration. Diarrhea categorized as mild: 2-3 loose stools in 24h; moderate: 4-5 loose stools in 24h; severe: 6 or more loose stools in 24h. Headache, fatigue, chills, new/worsened muscle pain and new/worsened joint pain were categorized as mild: didn't interfere with activity; moderate: some interference with activity; severe: prevented daily routine activity.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: Group 1: RSVpreF + qIRV | SSA: Group 2: qIRV
Number analyzed (Participants) | 125 | 125
Percentage of participants
  Fever: Mild | 4.0 [1.3 to 9.1] | 12.8 [7.5 to 20.0]
  Fever: Moderate | 6.4 [2.8 to 12.2] | 4.0 [1.3 to 9.1]
  Fever: Severe | 1.6 [0.2 to 5.7] | 5.6 [2.3 to 11.2]
  Fatigue: Mild | 20.8 [14.1 to 29.0] | 20.8 [14.1 to 29.0]
  Fatigue: Moderate | 30.4 [22.5 to 39.3] | 24.0 [16.8 to 32.5]
  Fatigue: Severe | 0.8 [0.0 to 4.4] | 4.0 [1.3 to 9.1]
  Headache: Mild | 24.0 [16.8 to 32.5] | 26.4 [18.9 to 35.0]
  Headache: Moderate | 24.8 [17.5 to 33.3] | 11.2 [6.3 to 18.1]
  Headache: Severe | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Vomiting: Mild | 1.6 [0.2 to 5.7] | 1.6 [0.2 to 5.7]
  Vomiting: Moderate | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Vomiting: Severe | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Nausea: Mild | 5.6 [2.3 to 11.2] | 5.6 [2.3 to 11.2]
  Nausea: Moderate | 2.4 [0.5 to 6.9] | 3.2 [0.9 to 8.0]
  Nausea: Severe | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  Diarrhea: Mild | 4.8 [1.8 to 10.2] | 4.0 [1.3 to 9.1]
  Diarrhea: Moderate | 1.6 [0.2 to 5.7] | 1.6 [0.2 to 5.7]
  Diarrhea: Severe | 0.8 [0.0 to 4.4] | 0 [0.0 to 2.9]
  Chills: Mild | 15.2 [9.4 to 22.7] | 20.8 [14.1 to 29.0]
  Chills: Moderate | 12.0 [6.9 to 19.0] | 11.2 [6.3 to 18.1]
  Chills: Severe | 0 [0.0 to 2.9] | 0 [0.0 to 2.9]
  New or worsened muscle pain: Mild | 17.6 [11.4 to 25.4] | 20.8 [14.1 to 29.0]
  New or worsened muscle pain: Moderate | 22.4 [15.4 to 30.7] | 15.2 [9.4 to 22.7]
  New or worsened muscle pain: Severe | 0 [0.0 to 2.9] | 1.6 [0.2 to 5.7]
  New or worsened joint pain: Mild | 11.2 [6.3 to 18.1] | 11.2 [6.3 to 18.1]
  New or worsened joint pain: Moderate | 14.4 [8.8 to 21.8] | 6.4 [2.8 to 12.2]
  New or worsened joint pain: Severe | 0 [0.0 to 2.9] | 0.8 [0.0 to 4.4]

5. Primary Outcome: SSA: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 2
Description: Systemic events included fever, fatigue, headache, vomiting, nausea, diarrhea, chills, new/worsened muscle pain and new/worsened joint pain. These were recorded by participants in an e-diary. Fever defined as oral temperature >=38.0 deg C and categorized as mild: >=38.0 to 38.4 deg C, moderate: >38.4 to 38.9 deg C, severe: >38.9 to 40.0 deg C. Vomiting categorized as mild: 1-2 times in 24h; moderate: >2 times in 24h; severe: required IV hydration. Diarrhea categorized as mild: 2-3 loose stools in 24h; moderate: 4-5 loose stools in 24h; severe: 6 or more loose stools in 24h. Headache, fatigue, chills, new/worsened muscle pain and new/worsened joint pain were categorized as mild: didn't interfere with activity; moderate: some interference with activity; severe: prevented daily routine activity.
Time Frame: SSA: From Day 1 to Day 7 after Vaccination 2 (1 Month after Vaccination 1)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: Group 1: Placebo | SSA: Group 2: RSVpreF
Number analyzed (Participants) | 121 | 115
Percentage of participants
  Fever: Mild | 0 [0.0 to 3.0] | 0.9 [0.0 to 4.7]
  Fever: Moderate | 0 [0.0 to 3.0] | 0.9 [0.0 to 4.7]
  Fever: Severe | 0 [0.0 to 3.0] | 0.9 [0.0 to 4.7]
  Fatigue: Mild | 7.4 [3.5 to 13.7] | 6.1 [2.5 to 12.1]
  Fatigue: Moderate | 3.3 [0.9 to 8.2] | 7.0 [3.1 to 13.2]
  Fatigue: Severe | 0 [0.0 to 3.0] | 1.7 [0.2 to 6.1]
  Headache: Mild | 10.7 [5.8 to 17.7] | 10.4 [5.5 to 17.5]
  Headache: Moderate | 5.8 [2.4 to 11.6] | 6.1 [2.5 to 12.1]
  Headache: Severe | 0 [0.0 to 3.0] | 0.9 [0.0 to 4.7]
  Vomiting: Mild | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Vomiting: Moderate | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Vomiting: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Nausea: Mild | 3.3 [0.9 to 8.2] | 1.7 [0.2 to 6.1]
  Nausea: Moderate | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Nausea: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Diarrhea: Mild | 5.0 [1.8 to 10.5] | 2.6 [0.5 to 7.4]
  Diarrhea: Moderate | 1.7 [0.2 to 5.8] | 0.9 [0.0 to 4.7]
  Diarrhea: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  Chills: Mild | 2.5 [0.5 to 7.1] | 3.5 [1.0 to 8.7]
  Chills: Moderate | 1.7 [0.2 to 5.8] | 2.6 [0.5 to 7.4]
  Chills: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  New or worsened muscle pain: Mild | 5.8 [2.4 to 11.6] | 4.3 [1.4 to 9.9]
  New or worsened muscle pain: Moderate | 1.7 [0.2 to 5.8] | 7.0 [3.1 to 13.2]
  New or worsened muscle pain: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]
  New or worsened joint pain: Mild | 4.1 [1.4 to 9.4] | 2.6 [0.5 to 7.4]
  New or worsened joint pain: Moderate | 1.7 [0.2 to 5.8] | 6.1 [2.5 to 12.1]
  New or worsened joint pain: Severe | 0 [0.0 to 3.0] | 0 [0.0 to 3.2]

6. Primary Outcome: SSB: Percentage of Participants With Systemic Events Within 7 Days After Vaccination
Description: as for outcome 5
Time Frame: SSB: From Day 1 to Day 7 After Vaccination
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 101 | 102
Percentage of participants
  Fever: Mild | 15.8 [9.3 to 24.4] | 10.8 [5.5 to 18.5]
  Fever: Moderate | 4.0 [1.1 to 9.8] | 2.0 [0.2 to 6.9]
  Fever: Severe | 2.0 [0.2 to 7.0] | 0 [0.0 to 3.6]
  Fatigue: Mild | 20.8 [13.4 to 30.0] | 28.4 [19.9 to 38.2]
  Fatigue: Moderate | 36.6 [27.3 to 46.8] | 26.5 [18.2 to 36.1]
  Fatigue: Severe | 0 [0.0 to 3.6] | 5.9 [2.2 to 12.4]
  Headache: Mild | 18.8 [11.7 to 27.8] | 26.5 [18.2 to 36.1]
  Headache: Moderate | 27.7 [19.3 to 37.5] | 15.7 [9.2 to 24.2]
  Headache: Severe | 0 [0.0 to 3.6] | 2.0 [0.2 to 6.9]
  Vomiting: Mild | 0 [0.0 to 3.6] | 2.0 [0.2 to 6.9]
  Vomiting: Moderate | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.3]
  Vomiting: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]
  Nausea: Mild | 5.0 [1.6 to 11.2] | 11.8 [6.2 to 19.6]
  Nausea: Moderate | 4.0 [1.1 to 9.8] | 2.9 [0.6 to 8.4]
  Nausea: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]
  Diarrhea: Mild | 9.9 [4.9 to 17.5] | 10.8 [5.5 to 18.5]
  Diarrhea: Moderate | 5.9 [2.2 to 12.5] | 2.9 [0.6 to 8.4]
  Diarrhea: Severe | 0 [0.0 to 3.6] | 0 [0.0 to 3.6]
  Chills: Mild | 15.8 [9.3 to 24.4] | 17.6 [10.8 to 26.4]
  Chills: Moderate | 24.8 [16.7 to 34.3] | 13.7 [7.7 to 22.0]
  Chills: Severe | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.3]
  New or worsened muscle pain: Mild | 18.8 [11.7 to 27.8] | 21.6 [14.0 to 30.8]
  New or worsened muscle pain: Moderate | 27.7 [19.3 to 37.5] | 22.5 [14.9 to 31.9]
  New or worsened muscle pain: Severe | 2.0 [0.2 to 7.0] | 1.0 [0.0 to 5.3]
  New or worsened joint pain: Mild | 14.9 [8.6 to 23.3] | 11.8 [6.2 to 19.6]
  New or worsened joint pain: Moderate | 20.8 [13.4 to 30.0] | 16.7 [10.0 to 25.3]
  New or worsened joint pain: Severe | 0 [0.0 to 3.6] | 1.0 [0.0 to 5.3]

7. Primary Outcome: SSA: Percentage of Participants Reporting Adverse Events (AEs) Within 1 Month After Vaccination 1
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were included.
Time Frame: SSA: Within 1 Month after Vaccination 1
Population: SSA: Safety population consisted of all enrolled participants who received the study intervention either in combination RSVpreF + qIRV, or as placebo, qIRV, or RSVpreF alone.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSA: Group 1: RSVpreF + qIRV | SSA: Group 2: qIRV
Number analyzed (Participants) | 125 | 126
Percentage of participants | 29.6 [21.8 to 38.4] | 33.3 [25.2 to 42.3]

8. Primary Outcome: SSA: Percentage of Participants Reporting AEs Within 1 Month After Vaccination 2
Description: as for outcome 7
Time Frame: SSA: Within 1 Month after Vaccination 2
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: Group 1: Placebo: Participants received 1 mL of combination of RSVpreF and qIRV intramuscularly on Day 1 [Vaccination 1].
- SSA: Group 2: RSVpreF: Participants received 1 mL of RSVpreF intramuscularly on 1 month apart Vaccination 1 [Vaccination 2].
Arm/Group | SSA: Group 1: Placebo | SSA: Group 2: RSVpreF
Number analyzed (Participants) | 121 | 116
Percentage of participants | 16.5 [10.4 to 24.4] | 13.8 [8.1 to 21.4]

9. Primary Outcome: SSB: Percentage of Participants Reporting AEs Throughout the Sub Study
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. Exact 2-sided 95% CI was based on the Clopper and Pearson method. Only AEs collected by non-systematic assessment (i.e. excluding local reactions and systemic events) were included.
Time Frame: SSB: From Day 1 of Vaccination up to 35 days of follow-up post Vaccination
Population: SSB: Safety population consisted of all enrolled participants who received the study intervention (0.5 mL or 1.0 mL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 101 | 102
Percentage of participants | 22.8 [15.0 to 32.2] | 33.3 [24.3 to 43.4]

10. Primary Outcome: SSA: Percentage of Participants Reporting Serious Adverse Events (SAEs) Throughout the Sub Study
Description: An SAE was defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria - resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect and was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic and other important medical event.
Time Frame: SSA: From Day 1 (Vaccination 1) up to 35 days of follow-up post Vaccination 2 (Maximum up to 70 days)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo: Participants aged >= 60 years received 1.0 mL combination of RSVpreF and qIRV intramuscularly on Day 1 [Vaccination 1]. After 1 month, placebo (0.9% normal saline for injection) [Vaccination 2] was administered intramuscularly. Participants were followed up to maximum of 35 days after Vaccination 2.
- SSA: Group 2: Sequential Administration qIRV/ RSVpreF: Participants aged >= 60 years received 1.0 mL of qIRV intramuscularly on Day 1 (Vaccination 1). After 1 month, RSVpreF (Vaccination 2) was administered intramuscularly. Participants were followed up to maximum of 35 days after Vaccination 2.
Arm/Group | SSA: Group 1: Combination (RSVpreF + qIRV)/ Placebo | SSA: Group 2: Sequential Administration qIRV/ RSVpreF
Number analyzed (Participants) | 125 | 126
Percentage of participants | 0 [0.0 to 2.9] | 2.4 [0.5 to 6.8]

11. Primary Outcome: SSB: Percentage of Participants Reporting SAEs Throughout the Sub Study
Description: as for outcome 10
Time Frame: SSB: From Day 1 of Vaccination up to 35 days of follow-up post Vaccination (Maximum up to 36 days)
Population: SSB: Safety population consisted of all enrolled participants who received the study intervention (0.5 mL or 1.0 mL).
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 101 | 102
Percentage of participants | 2.0 [0.2 to 7.0] | 0 [0.0 to 3.6]

12. Primary Outcome: SSA: Geometric Mean Titer (GMT) and Geometric Mean Ratio (GMR) of Neutralizing Titers (NT) for Each RSV Subgroup (A or B) 1 Month After Vaccination With Combination RSVpreF + qIRV (Group 1) and RSVpreF Alone (Group 2)
Description: GMTs and associated 2-sided 95% CIs are reported as descriptive data. GMRs and associated 2-sided 95% CIs are reported in statistical analysis section of this outcome measure. GMR was the ratio of RSV subgroup A (RSV A) or RSV subgroup B (RSV B) neutralizing GMTs in the combination RSVpreF + qIRV group to that in the sequential-administration RSVpreF group.
Time Frame: SSA- For Group 1: 1 Month after Vaccination 1 (Day 1); For Group 2: 1 Month after Vaccination 2 (1 Month after Vaccination 1)
Population: Evaluable RSV immunogenicity population: all eligible participants who received the study intervention to which they were randomized, had the 1 month postvaccination blood collection within 27 to 42 days after vaccination, had at least 1 valid and determinate RSV NT result at the 1-month postvaccination blood collection, and had no major protocol violations from randomization through the 1 month postvaccination blood collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Groups:
- SSA: Group 1: Combination RSVpreF + qIRV: Participants received 1 mL combination of RSVpreF and qIRV intramuscularly on Day 1 [Vaccination 1].
- SSA: Group 2: Sequential Administration RSVpreF Alone: Participants received 1 mL of RSVpreF intramuscularly on 1 month after Vaccination 1 [Vaccination 2]
Arm/Group | SSA: Group 1: Combination RSVpreF + qIRV | SSA: Group 2: Sequential Administration RSVpreF Alone
Number analyzed (Participants) | 119 | 112
Titer
  NT: RSV A | 16553 [14120.9 to 19403.1] | 19740 [16555.5 to 23536.4]
  NT: RSV B | 11795 [9961.1 to 13966.7] | 14959 [12408.8 to 18032.4]
Statistical Analysis 1: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for RSV A: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; GMR = 0.84, 95% CI 2-sided [0.662 to 1.062]
Statistical Analysis 2: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for RSV B: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; GMR = 0.79, 95% CI 2-sided [0.614 to 1.013]

13. Primary Outcome: SSA: GMT and GMR of Strain-Specific Hemagglutination Inhibition (HAI) Titers For 1 Month After Vaccination With Combination RSVpreF + qIRV (Group 1) and qIRV Alone (Group 2)
Description: GMTs and associated 2-sided 95% CIs are reported as descriptive data. GMRs and associated 2-sided 95% CIs are reported in statistical analysis section of this outcome measure. GMR was the ratio of each strain neutralizing GMTs in the combination RSVpreF + qIRV group to that in the sequential-administration RSVpreF group. The analysis was performed on the influenza strains: H1N1 A/Sydney, H3N2 A/Darwin, B/Austria, and B/Phuket.
Time Frame: as for outcome 12
Population: Evaluable HAI immunogenicity population: all eligible participants who received the study intervention to which they were randomized, and had the 1month postvaccination blood collection for HAI assay within 27-42 days after vaccination, had at least 1 valid and determinate HAI result at 1 month postvaccination blood collection, had no major protocol violations from randomization through 1 month postvaccination blood collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSA: Group 1: Combination RSVpreF + qIRV | SSA: Group 2: Sequential Administration RSVpreF Alone
Number analyzed (Participants) | 119 | 112
Titer
  HAI: H1N1 A/Wisconsin | 194 [164.3 to 227.9] | 238 [196.5 to 288.7]
  HAI: H3N2 A/Darwin | 161 [136.9 to 189.9] | 219 [178.1 to 269.0]
  HAI: B/Austria | 53 [44.6 to 62.1] | 56 [47.7 to 66.3]
  HAI: B/Phuket | 22 [18.5 to 26.4] | 24 [20.2 to 29.1]
Statistical Analysis 1: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for HAI: H1N1 A/Wisconsin: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; GMR = 0.81, 95% CI 2-sided [0.632 to 1.044]
Statistical Analysis 2: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for HAI: H3N2 A/Darwin: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; Geometric Mean Ratio = 0.74, 95% CI 2-sided [0.567 to 0.957]
Statistical Analysis 3: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for HAI: B/Austria: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; GMR = 0.94, 95% CI 2-sided [0.741 to 1.181]
Statistical Analysis 4: Comparison: SSA: Group 1: Combination RSVpreF + qIRV vs SSA: Group 2: Sequential Administration RSVpreF Alone; GMR for HAI: B/Phuket: RSVpreF + qIRV combination to RSVpreF alone; Test type: Other; GMR = 0.91, 95% CI 2-sided [0.707 to 1.174]

14. Secondary Outcome: SSB: GMT and GMR of NT for Each RSV A or RSV B 1 Month After Vaccination
Description: GMTs and associated 2-sided 95% CIs are reported as descriptive data. GMRs and associated 2-sided 95% CIs are reported in statistical analysis section of this outcome measure. GMR was the ratio of RSV A or RSV B neutralizing GMTs in the combination of 1 mL RSVpreF + qIRV (group 1) and 0.5 ml of RSVpreF + qIRV (group 2)
Time Frame: SSB: At 1 Month after Vaccination (Day 1)
Population: Evaluable RSV immunogenicity population: all eligible participants who received the study intervention to which they were randomized, had the 1-month postvaccination blood collection within 27 to 42 days after vaccination, had at least 1 valid and determinate RSV NT result at the 1 month postvaccination blood collection, and had no major protocol violations from randomization through the 1 month postvaccination blood collection.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 100 | 99
Titer
  NT: RSV A | 32044 [26676.5 to 38492.2] | 30575 [25922.1 to 36062.4]
  NT: RSV B | 30364 [25533.4 to 36108.2] | 28614 [24113.5 to 33954.8]
Statistical Analysis 1: Comparison: SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation vs SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for RSV A: RSVpreF + qIRV 1.0 mL (Group 1) combination to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; Geometric Mean Ratio = 1.05, 95% CI 2-sided [0.820 to 1.339]
Statistical Analysis 2: Comparison: SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation vs SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for RSV B: RSVpreF + qIRV 1.0 mL (Group 1) to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; Geometric Mean Ratio = 1.06, 95% CI 2-sided [0.833 to 1.352]

15. Secondary Outcome: SSB: GMTs of Strain-Specific Hemagglutination Inhibition (HAI) at 1 Month After Vaccination
Description: GMTs and associated 2-sided 95% CIs are reported as descriptive data. GMRs and associated 2-sided 95% CIs are reported in statistical analysis section of this outcome measure. GMR was the ratio of each strain neutralizing GMTs to the combination of 1 mL RSVpreF + qIRV (Group 1) and 0.5 ml of RSVpreF + qIRV (Group 2). The analysis was performed on the influenza strains: H1N1 A/Sydney, H3N2 A/Darwin, B/Austria, and B/Phuket.
Time Frame: SSB: At 1 Month after Vaccination (Day 1)
Population: Evaluable HAI immunogenicity population: all eligible participants who received the study intervention to which they were randomized, and had the 1month postvaccination blood collection for HAI assay within 27-42 days after vaccination,had atleast 1 valid and determinate HAI result at 1 month postvaccination blood collection,had no major protocol violations from randomization through 1 month postvaccination blood collection. 'Number Analyzed'=participants evaluable for specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
Number analyzed (Participants) | 100 | 99
Titer
  HAI: H1N1 A/Sydney | 257 [212.6 to 311.8] | 217 [170.2 to 275.8]
  HAI: H3N2 A/Darwin: number analyzed (Participants) | 99 | 98
  HAI: H3N2 A/Darwin | 259 [216.4 to 310.8] | 229 [188.7 to 279.0]
  HAI: B/Austria | 58 [49.0 to 69.0] | 54 [45.0 to 64.1]
  HAI: B/Phuket | 32 [27.0 to 38.6] | 29 [25.1 to 34.4]
Statistical Analysis 1: Comparison: SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for HAI: H1N1 A/Sydney: RSVpreF + qIRV 1.0 mL (Group 1) to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; GMR = 1.19, 95% CI 2-sided [0.875 to 1.614]
Statistical Analysis 2: Comparison: SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation vs SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for HAI: H3N2 A/Darwin: RSVpreF + qIRV 1.0 mL (Group 1) to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; Geometric Mean Ratio = 1.13, 95% CI 2-sided [0.867 to 1.473]
Statistical Analysis 3: Comparison: SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation vs SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for HAI: B/Austria: RSVpreF + qIRV 1.0 mL (Group 1) to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; Geometric Mean Ratio = 1.08, 95% CI 2-sided [0.849 to 1.383]
Statistical Analysis 4: Comparison: SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation vs SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation; GMR for HAI: B/Phuket: RSVpreF + qIRV 1.0 mL (Group 1) to RSVpreF + qIRV 0.5 mL (Group 2); Test type: Other; Geometric Mean Ratio = 1.10, 95% CI 2-sided [0.866 to 1.392]

ADVERSE EVENTS:
Time Frame: Local reactions/systemic events (systematic assessment): Day 1 up to Day 7 after each Vaccination; AEs (non-systematic assessment): SSA- Day 1 up to 35 days after Vaccination 2 (Maximum up to approximately 70 days) and SSB- Day 1 up to 35 days after Vaccination (Maximum up to approximately 36 days)
Description: Same event may appear as both SAE and non-SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. MedDRA versions used were v26.0 for SSA and v26.1 for SSB.
Groups:
- SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation: Participants aged >=50 years were randomized to receive 1.0 mL of combination of RSVpreF and qIRV intramuscularly on Day 1.
- SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation: Participants aged >=50 years were randomized to receive 0.5 mL of combination of RSVpreF and qIRV intramuscularly on Day 1.
Arm/Group | SSA: Group 1: RSVpreF + qIRV | SSA: Group 1: Placebo | SSA: Group 2: qIRV | SSA: Group 2: RSVpreF | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation
All-Cause Mortality (participants affected / at risk) | 0/125 | 0/121 | 0/126 | 1/116 | 0/101 | 0/102
Serious Adverse Events (participants affected / at risk) | 0/125 | 0/121 | 1/126 | 1/116 | 2/101 | 0/102
Other Adverse Events (participants affected / at risk) | 117/125 | 50/121 | 117/126 | 43/116 | 91/101 | 96/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SSA: Group 1: RSVpreF + qIRV (N=125) | SSA: Group 1: Placebo (N=121) | SSA: Group 2: qIRV (N=126) | SSA: Group 2: RSVpreF (N=116) | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation (N=101) | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation (N=102)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | SSA: Group 1: RSVpreF + qIRV (N=125) | SSA: Group 1: Placebo (N=121) | SSA: Group 2: qIRV (N=126) | SSA: Group 2: RSVpreF (N=116) | SSB: Group 1: RSVpreF + qIRV 1.0 mL Formulation (N=101) | SSB: Group 2: RSVpreF + qIRV 0.5 mL Formulation (N=102)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Cardiac septal hypertrophy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Dilated cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Left atrial dilatation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Axillary pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 2 | 3 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Influenza like illness (General disorders) | 2 | 3 | 2 | 0 | 2 | 9 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site bruising (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site erythema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site lymphadenopathy (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Vaccination site papule (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Chronic gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Coeliac disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Odynophagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Atypical pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Bronchitis (Infections and infestations) | 4 | 0 | 0 | 0 | 2 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Conjunctivitis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 1 | 2 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 2 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Buttock injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 1 | 1 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Joint injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Troponin T increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 2 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Dizziness (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Tension headache (Nervous system disorders) | 1 | 1 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Trigeminal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Renal disorder (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Catarrh (Respiratory, thoracic and mediastinal disorders) | 15 | 6 | 13 | 4 | 4 | 12 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Hypertension (Vascular disorders) | 2 | 0 | 6 | 0 | 2 | 2 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Chills (CHILLS) (General disorders) | 34 | 5 | 40/125 | 7/115 | 41 | 33 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Fatigue (FATIGUE) (General disorders) | 65 | 13 | 61/125 | 17/115 | 58 | 62 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site erythema (REDNESS) (General disorders) | 9 | 0 | 11/125 | 0/115 | 2 | 6 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site pain (PAIN AT THE INJECTION SITE) (General disorders) | 88 | 4 | 103/125 | 10/115 | 76 | 80 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Injection site swelling (SWELLING) (General disorders) | 12 | 1 | 21/125 | 1/115 | 10 | 14 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Pyrexia (FEVER) (General disorders) | 15 | 0 | 28/125 | 3/115 | 22 | 13 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Diarrhoea (DIARRHEA) (Gastrointestinal disorders) | 9 | 8 | 7/125 | 4/115 | 16 | 14 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Nausea (NAUSEA) (Gastrointestinal disorders) | 10 | 4 | 11/125 | 2/115 | 9 | 15 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Vomiting (VOMITING) (Gastrointestinal disorders) | 2 | 0 | 2/125 | 0/115 | 0 | 3 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Arthralgia (NEW OR WORSENED JOINT PAIN) (Musculoskeletal and connective tissue disorders) | 32 | 7 | 23/125 | 10/115 | 36 | 30 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Myalgia (NEW OR WORSENED MUSCLE PAIN) (Musculoskeletal and connective tissue disorders) | 50 | 9 | 47/125 | 13/115 | 49 | 46 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB
Headache (HEADACHE) (Nervous system disorders) | 61 | 20 | 47/125 | 20/115 | 47 | 45 — MedDRA v26.0 for SSA, MedDRA v26.1 for SSB

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05788237/Prot_000.pdf
  • Statistical Analysis Plan (2023-07-14): https://cdn.clinicaltrials.gov/large-docs/37/NCT05788237/SAP_001.pdf